CLINICAL TRIAL: NCT01663415
Title: A Phase 2, Multicenter, Single-arm Study to Evaluate the Safety and Efficacy of Enzalutamide in Chemotherapy-Naïve, Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Enzalutamide in Chemotherapy-Naïve, Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision was made to not initiate this study.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-UC-0001
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: MDV3100; prostate; cancer; enzalutamide
MeSH Terms: conditions — Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Experimental)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — oral
  Other Names: MDV3100

SUMMARY:
The purpose of this study is to investigate radiographic progression-free survival (PFS) of enzalutamide in chemotherapy-naïve patients with progressive metastatic castration-resistant prostate cancer who have symptomatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Progressive prostate cancer while on androgen deprivation therapy
* Castrate testosterone level
* Maintenance of surgical or medical castration for duration of study
* Radiographically visible metastatic disease
* Symptomatic from prostate cancer
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Life expectancy >=6 months

Exclusion Criteria:

* Brain metastases or leptomeningeal disease
* Prior cytotoxic chemotherapy for prostate cancer
* Prior use of ketoconazole or abiraterone acetate or other investigational agent that blocks androgen synthesis or targets androgen receptor
* History of seizure or condition that may predispose to seizure
* History of loss of consciousness or transient ischemic attack within 12 months
* Clinically significant cardiovascular disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression free survival (PFS) | 26 months
  Time from first dose on Day 1 to the first objective evidence of radiographic progression or death due to any cause (whichever occurs first). Radiographic disease progression is defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Prostate Cancer Clinical Trials Working Group 2 (PCWG2).

SECONDARY OUTCOMES:
Overall survival | 26 months
  Time from first dose on Day 1 to death due to any cause
Time to PSA progression | 26 months
  Time from first dose on Day 1 to first observation of PSA progression
Change from baseline to last post baseline measurement Quality of life score using Functional Assessment of Cancer Therapy-Prostate (FACT-P) | Baseline and 26 months
  The FACT-P quality of life questionnaire is a multi-dimensional, self-reported quality of life instrument specifically designed for use with prostate cancer patients
Change from baseline to last post baseline measurement Quality of Life score using European Quality of Life 5-Domain Scale (EQ-5D) | Baseline and 26 months
  EQ-5D is a standardized instrument for use as a measure of health outcome. It provides a simple descriptive profile and a single index value for health status and is designed for self-completion by respondents
Change from baseline to last post baseline measurement Pain Assessments (Brief Pain Inventory - Short Form) | Baseline and 26 months
  Brief Pain Inventory is a validated instrument that is a subject self-rating scale assessing level of pain, effect of the pain on activities of daily living, and analgesic use
Safety assessed by recording of adverse events, safety laboratory evaluations, vital signs and electrocardiograms (ECGs) | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development